CLINICAL TRIAL: NCT06264492
Title: Deciphering Patient Participation: Insights From Observational Data in Scleroderma Clinical Trials
Brief Title: Delving Into Participation Trends of Scleroderma Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 55777205
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Scleroderma
Keywords: scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Typically, specific demographic subsets tend to exhibit greater engagement in medical research. Nonetheless, there is insufficient research elucidating the trial characteristics influencing the participation of these particular demographics.

The study will analyze data from diverse demographic viewpoints to uncover recurring trends that could provide valuable insights for future patients with scleroderma.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with scleroderma
* Patient has self-identified as planning to enroll in an observational clinical trial
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient is pregnant
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with scleroderma who are actively considering participation in a clinical trial for this ailment, but have not yet concluded the enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients in clinical research for scleroderma | 3 months
Number of scleroderma study participants who stay committed until clinical study wraps up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Careta MF, Leite Cda C, Cresta F, Albino J, Tsunami M, Romiti R. Prospective study to evaluate the clinical and radiological outcome of patients with scleroderma of the face. Autoimmun Rev. 2013 Sep;12(11):1064-9. doi: 10.1016/j.autrev.2013.05.005. Epub 2013 Jun 19. PMID 23791631
- [Background] Harb S, Pelaez S, Carrier ME, Kwakkenbos L, Bartlett SJ, Hudson M, Mouthon L, Sauve M, Welling J, Shrier I, Thombs BD; SPIN Physical Activity Enhancement Patient Advisory Team and SPIN Investigators. Barriers and Facilitators to Physical Activity for People With Scleroderma: A Scleroderma Patient-Centered Intervention Network Cohort Study. Arthritis Care Res (Hoboken). 2022 Aug;74(8):1300-1310. doi: 10.1002/acr.24567. Epub 2022 May 11. PMID 33527717
- [Background] Li SC. Treatment of juvenile localized scleroderma: current recommendations, response factors, and potential alternative treatments. Curr Opin Rheumatol. 2022 Sep 1;34(5):245-254. doi: 10.1097/BOR.0000000000000886. PMID 35880663

DOCUMENTS (1):
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT06264492/ICF_000.pdf